CLINICAL TRIAL: NCT05605223
Title: Study of Acute Autoimmune Encephalitis With Positive Antibodies in Eastern France Between 2006 and 2018
Brief Title: Study of Acute Autoimmune Encephalitis With Positive Antibodies in Eastern France
Acronym: Encephalitis
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7415
Record Dates: First submitted 2022-10-28; First posted 2022-11-04 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Acute Autoimmune Encephalitis
Keywords: Acute autoimmune encephalitis; encephalitis; autoimmune encephalitis
MeSH Terms: conditions — Encephalitis; Autoimmune Diseases of the Nervous System

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The number of acute encephalitides diagnosed each year is gradually increasing, reaching approximately 5 to 10/100,000 per year; more than 50% of etiologies currently remain unknown. The majority of them are acute encephalitis of infectious origin, but it is estimated that 20% of encephalitis in northern Europe is related to an autoimmune mechanism with the majority of encephalitis with anti-NMDA Ac discovered recently in 2007. The study of a large American encephalitis cohort showed a death rate of 3% to 7% in cases of autoimmune encephalitis. Furthermore, delay in the initiation of effective treatment (tumor removal or immunotherapy) beyond 4 weeks is associated with a poor prognosis at 1 year.

It is therefore necessary to better understand the signs of autoimmune encephalitis in order to recognize the disease quickly and to start a treatment quickly; in order to improve the management and the prognosis of these children.

ELIGIBILITY:
Inclusion criteria:

* Age between 0 and 17 years at diagnosis
* Patient diagnosed between 01/01/2006 and 31/12/2018 with autoimmune encephalitis in one of the participating university hospitals (Besançon, Nancy, Strasbourg, Reims and Dijon)
* Presence of clinical criteria of clinical and/or radiographic encephalitis
* Presence of one or more antibodies in the blood or CSF
* Parental authority holders and their child of childbearing age having given their consent for the use of the child's data for this research

Exclusion criteria:

* Refusal to participate in the study
* Absence of consultation at any of the study centers
* Absence of clinical and/or radiographic criteria for encephalitis.
* Absence of antibodies found in blood or CSF

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Minor subject (≤17 years) diagnosed between 01/01/2006 and 31/12/2018 with autoimmune encephalitis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2019-10-26 (Actual); Study Completion 2019-12-26 (Actual)

PRIMARY OUTCOMES:
Retrospective description of autoimmune encephalitis in children | Files analysed retrospectively from January 01, 2006 to December 31, 2018 will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pédiatrie 1 - CHU de Strasbourg - France, Strasbourg, France